CLINICAL TRIAL: NCT01327703
Title: An Open-label, Multicenter, Randomized, Cross-over Study to Compare the Safety and Efficacy of PANZYTRAT® 25,000 to KREON® 25,000 in the Control of Steatorrhea in Subjects Aged 7 Years and Older With Cystic Fibrosis (CF) and Exocrine Pancreatic Insufficiency (EPI)
Brief Title: Control of Steatorrhea in Participants With Cystic Fibrosis and Exocrine Pancreatic Insufficiency
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MA-PA25CF10-01; 2010-019267-11 (EudraCT Number)
Record Dates: First submitted 2011-03-28; First posted 2011-04-04 (Estimated); Results first posted 2014-04-10 (Estimated); Last update posted 2014-04-10 (Estimated); Status verified 2014-03

CONDITIONS: Exocrine Pancreatic Insufficiency; Cystic Fibrosis
Keywords: Exocrine Pancreatic Insufficiency; Cystic Fibrosis; Steatorrhea; Malabsorption; Malnutrition
MeSH Terms: conditions — Exocrine Pancreatic Insufficiency; Cystic Fibrosis; Steatorrhea; Malabsorption Syndromes; Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Panzytrat® 25,000 (Experimental)
  Interventions: Drug: Panzytrat® 25,000
- Kreon® 25,000 (Active Comparator)
  Interventions: Drug: Kreon® 25,000

INTERVENTIONS:
Drug: Panzytrat® 25,000 — Panzytrat® 25,000 capsule will be given orally daily at a stabilized dose, as per investigator's discretion, for 14 days. Stabilized dose for a participant will be the optimal dose determined during a qualification phase that precedes the first treatment period and will be based upon the participant's usual lipase and lipid intake. Total dose will not exceed 10,000 European Pharmacopoeia (Ph.Eur.) units lipase/kilogram (kg) body weight/day in either first treatment period or second treatment period.
  Arms: Panzytrat® 25,000
Drug: Kreon® 25,000 — Kreon® 25,000 capsule will be given orally daily at a stabilized dose, as per investigator's discretion, for 14 days. Stabilized dose for a participant will be the optimal dose determined during a qualification phase that precedes the first treatment period and will be based upon the participant's usual lipase and lipid intake. Total dose will not exceed 10,000 Ph.Eur. units lipase/kg body weight/day in either first treatment period or second treatment period.
  Arms: Kreon® 25,000

SUMMARY:
This study by Aptalis (formerly Axcan) assesses the efficacy and safety of Panzytrat® 25,000 compared to Kreon® 25,000 in the control of steatorrhea in participants with cystic fibrosis (CF) and exocrine pancreatic insufficiency (EPI).

DETAILED DESCRIPTION:
This is an open-label, Phase IV, multicenter, randomized, two-period cross-over study to compare the efficacy and safety of Panzytrat® 25,000 to Kreon® 25,000 in participants aged 7 years and older suffering from CF and EPI. The study consists of a qualification phase (5 to 15 days); two treatment periods of 14 days each (plus a 3-day window if needed) and a 3-day stool collection will be performed from Days 12 to 15.

A safety follow-up phone call will be arranged 7-10 days after completion of the treatment phase or after an early discontinuation.

ELIGIBILITY:
Inclusion Criteria:

* Participant or his/her legal representative signed informed consent form (ICF) prior to starting any study procedures
* Participant with clinical diagnosis of CF based on one or more typical clinical features of CF phenotype, in addition to one of the following: a genotype that documents the presence of 2 CF-causing mutation, or a sweat chloride test greater than or equal to 60 millimole per liter (mmol/L) by quantitative pilocarpine iontophoresis on two separate occasions
* Participant with severe EPI confirmed by enzyme-linked immunosorbent assay (ELISA) measurement of fecal elastase-1 (FE-1)
* Male or female participant aged 7 years or older
* Participant currently receiving and has received a stable dose of lipase with either Panzytrat® 25,000 or Kreon® 25,000 for at least 30 days prior to ICF signature
* Participant generally in good health, except for the underlying symptoms associated with CF and EPI, and is clinically stable (no change in the last 30 days of physical examination) as evidenced by medical and medication histories, physical examination including vital signs during screening and laboratory tests
* Participant able to maintain a CF standardized diet with a lipid content customized to his/her needs during the study according to the qualification phase diary
* Women of childbearing potential must have a negative pregnancy test at study entry and must use a medically acceptable contraceptive method for the duration of the study

Exclusion Criteria:

* Participant with known contraindication, sensitivity or hypersensitivity to Panzytrat® 25,000 or Kreon® 25,000, or to any porcine protein
* Participant who recently received treatment of an emergent acute infection with oral or intravenous (IV) antibiotics that was not stopped at least 14 days prior to randomization
* Participant with chronic use of narcotics that were not stopped at least 7 days prior to the qualification visit
* Participant using of any prohibited medications or products listed in the prohibited medication section of the protocol
* Participant with acute pancreatitis or exacerbation of chronic pancreatic disease
* Participant with history of significant bowel resection that could impair fat absorption
* Participant with any condition known to increase fecal fat loss including but not limited to: celiac disease, Crohn's disease, tropical sprue, bacterial bowel infection, liver disease, lactose intolerance, pseudomembranous colitis, biliary and pancreatic cancer, radiation enteritis, Whipple's disease, Whipple's procedure, etc
* Participant with any significant gastrointestinal dysmotility disorders
* Participant with chronic abdominal pain or severe abdominal pain at study entry
* Participant using enteral tube feeding over day and night
* Participant with history or presence of clinically significant portal hypertension
* Participant with history or presence of complete distal intestinal obstruction syndrome (DIOS) in the past 6 months, or 2 or more episodes of DIOS in the past year
* Participant with poorly controlled diabetes as per the investigator's opinion
* Female participants who are pregnant or breastfeeding
* Participant with any condition or history of any illness, or pre-study laboratory abnormality which, in the opinion of the investigator or sponsor, might put the participant at risk, prevent the participant from completing the study, or otherwise affect the outcome of the study
* Participant using any investigational drug within 30 days prior to the date of signature of the ICF

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2011-04; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aptalis Medical Information, Study Director — Forest Laboratories
Locations (13):
- Germany (6):
  - Klinikum-Bochum, Bochum
  - Universitätsklinikum Carl Gustav Carus, Dresden
  - Universitaetsklinikum Erlangen, Erlangen
  - Jena University Hospital, Universitaetsklinikum Jena, Jena
  - Klinikum der Universitat Munchen Medizinische Klinik-Innenstadt, München
  - University Children's Clinic Tubingen, Tübingen
- Poland (7):
  - Specjalistyczny Zespół Opieki Zdrowotnej nad Matką i Dzieckiem Poradnia Leczenia Mukowiscydozy, Gdansk
  - Wojewodzki Specjalistityczny Szpital Dziect Im Sw Ludwika, Krakow
  - Dziecięcy Szpital Kliniczny im. Prof. Antoniego Gębali, Lublin
  - Szpital Kliniczny im Karola Jonschera, Poznan
  - NZOZ Sanatorium Cassia Villa Medica, Rabka-Zdrój
  - NZOZ Podkarpacki Osrodek Pulmonologii i Alergologii, Rzeszów
  - Children's Health Memorial Institute, Warsaw

RESULTS

PARTICIPANT FLOW:
Groups:
- Panzytrat® First, Then Kreon®: Panzytrat® 25,000 capsule orally daily at a stabilized dose, as per investigator's discretion, for 14 days in first treatment period followed by Kreon® 25,000 capsule orally daily at a stabilized dose, as per investigator's discretion, for 14 days in second treatment period. Stabilized dose for a participant was the optimal dose determined during a qualification phase that preceded the first treatment period and was based upon the participant's usual lipase and lipid intake and total dose was not to exceed 10,000 European Pharmacopoeia (Ph.Eur.) units lipase/kilogram (kg) body weight/day.
- Kreon® First, Then Panzytrat®: Kreon® 25,000 capsule orally daily at a stabilized dose, as per investigator's discretion, for 14 days in first treatment period followed by Panzytrat® 25,000 capsule orally daily at a stabilized dose, as per investigator's discretion, for 14 days in second treatment period. Stabilized dose for a participant was the optimal dose determined during a qualification phase that preceded the first treatment period and was based upon the participant's usual lipase and lipid intake and total dose was not to exceed 10,000 Ph.Eur. units lipase/kg body weight/day.
Period: First Treatment Period
Arm/Group | Panzytrat® First, Then Kreon® | Kreon® First, Then Panzytrat®
Started | 42 | 45
Completed | 42 | 45
Not Completed | 0 | 0
Period: Second Treatment Period
Arm/Group | Panzytrat® First, Then Kreon® | Kreon® First, Then Panzytrat®
Started | 40 (Two participants discontinued between first and second treatment periods due to adverse event.) | 44 (One participant discontinued between first and second treatment periods due to adverse event.)
Completed | 39 | 42
Not Completed | 1 | 2
Not completed — Adverse Event | 1 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all randomized participants.
Groups:
- Entire Study Population: Includes randomized participants who received Panzytrat® 25,000 first and Kreon® 25,000 first.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 87
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.6 (6.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 53
Nutritional status as assessed by Vitamin A and E level [Mean (Standard Deviation); unit: micromole/liter (mcmol/L)] — Nutritional status was assessed by determining Vitamin A and E (Alpha-Tocopherol and Beta-Gamma-Tocopherol) level. Here, 'n' signifies number of participants who were evaluable for the specific categories of this baseline characteristic.
  micromole/liter (mcmol/L)
    Vitamin A (n=87) | 1.403 (0.5329)
    Vitamin E (Alpha-Tocopherol) (n=87) | 18.554 (8.9713)
    Vitamin E (Beta-Gamma-Tocopherol) (n=83) | 1.231 (2.0781)
Nutritional status as assessed by Vitamin D level [Mean (Standard Deviation); unit: nanomole/L (nmol/L)] — Nutritional status was assessed by determining Vitamin D level. Number of participants who were evaluable for Vitamin D level was 86.
  nanomole/L (nmol/L) | 55.4 (33.24)

OUTCOME MEASURES:

1. Primary Outcome: Percent Coefficient of Fat Absorption (CFA)
Description: Percent CFA was calculated as ([fat intake - fat excretion]/fat intake)*100, determined in the stools which were collected over a 3-day period (Day 12 to morning of Day 15) during each treatment period. Least squares mean percent (%) CFA was calculated for Day 12 to Day 15 in first and second treatment periods. Percent CFA was based on log transformed data.
Time Frame: Day 12 up to Day 15 in first and second treatment periods
Population: Per protocol population included all randomized participants who completed both treatment periods and had all bowel movements appropriately collected with no major protocol violations/deviations or other events considered to potentially bias the study evaluations.
Measure: Least Squares Mean (Standard Error); unit: percent CFA
Groups:
- Panzytrat®: Panzytrat® 25,000 capsule orally daily at a stabilized dose, as per investigator's discretion, for 14 days in either first treatment period or second treatment period.
- Kreon®: Kreon® 25,000 capsule orally daily at a stabilized dose, as per investigator's discretion, for 14 days in either first treatment period or second treatment period.
Arm/Group | Panzytrat® | Kreon®
Number analyzed (Participants) | 38 | 38
percent CFA | 78.27 (1.033) | 80.35 (1.033)
Statistical Analysis 1: Comparison: Panzytrat® vs Kreon®; Mixed model analysis method was used for comparison using log-transformed percent CFA as the response variable, fixed effect factors for treatment, period, treatment sequence and pooled site and participant within treatment sequence as a random effect; Test type: Non-Inferiority or Equivalence — Non-inferiority was declared if the lower bound of the 2-sided 95% confidence interval (CI) of Panzytrat® versus Kreon® exceeded -10%; p = 0.4590, Mixed Models Analysis — As there was only a single pre-specified primary analysis, there was no adjustment for multiplicity; Treatment difference = -2.08, 95% CI 2-sided [-7.23 to 4.02]

2. Secondary Outcome: Mean Daily Number of Stools
Description: Mean daily number of stools of each participant was calculated from frequency of stools by the participant per day. Mean daily number of stools during the collection period (Day 12 to Day 15 in first and second treatment periods) for total participants was summarized.
Time Frame: Day 12 up to Day 15 in first and second treatment periods
Population: Intent-to-treat (ITT) population included all randomized participants. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: stools per day
Arm/Group | Panzytrat® | Kreon®
Number analyzed (Participants) | 85 | 84
stools per day | 4.5 (2.43) | 4.2 (2.14)

3. Secondary Outcome: Percentage of Stools With Normal Consistency
Description: Normal consistency of stool was defined as formed hard, normal or soft stool and abnormal consistency was defined as loose and unformed, liquid stool and diarrhea. Percentage of stools with normal consistency of each participant was calculated as the number of stools with normal consistency relative to the total number of stools during the collection period. Mean percentage of stool with normal consistency during the collection period (Day 12 to Day 15 in first and second treatment periods) for total participants was summarized.
Time Frame: Day 12 up to Day 15 in first and second treatment periods
Population: ITT population included all randomized participants. Here, 'N' (number of participants analyzed) specify signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: percentage of stools
Arm/Group | Panzytrat® | Kreon®
Number analyzed (Participants) | 83 | 83
percentage of stools | 0.644 (0.3442) | 0.635 (0.3517)

4. Secondary Outcome: Total Weight of Stools
Description: Mean total weight of stools was calculated for Day 12 to Day 15 in first and second treatment periods.
Time Frame: Day 12 up to Day 15 in first and second treatment periods
Population: ITT population included all randomized participants. Here, 'N' (number of participants analyzed) signifies those participants who had 1 or more bowel movements over the 72-hour collection period.
Measure: Mean (Standard Deviation); unit: gram
Arm/Group | Panzytrat® | Kreon®
Number analyzed (Participants) | 85 | 84
gram | 521.6 (301.95) | 484.0 (326.81)

5. Secondary Outcome: Mean Weight Per Stool Sample
Description: Mean weight per stool sample was calculated for Day 12 to Day 15 in first and second treatment periods.
Time Frame: Day 12 up to Day 15 in first and second treatment periods
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: gram
Arm/Group | Panzytrat® | Kreon®
Number analyzed (Participants) | 83 | 82
gram | 131.7 (79.67) | 124.0 (81.71)

6. Secondary Outcome: Relative Frequency of Days With Abdominal Symptoms
Description: Abdominal symptoms included abdominal pain and flatulence. Symptoms were classified by severity as mild (no impairment of daily activities), moderate (slight impairment of daily activities), or severe (unable to perform daily activities). For each type of abdominal symptom, the relative frequency of days with the symptom for each participant in a treatment period was calculated as the number of days in which the symptom was reported divided by the total number of days in which the abdominal symptom case report form (CRF) was completed. Mean relative frequency of days with abdominal symptoms was calculated during each treatment period (Day 1 to Day 15).
Time Frame: Day 1 up to Day 15 in first and second treatment periods
Population: ITT population included all randomized participants. Here, 'N' specifies number of participants who were evaluable for this outcome measure and 'n' specifies the number of participants with at least one report of the symptom at that severity level during a treatment period.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Panzytrat® | Kreon®
Number analyzed (Participants) | 86 | 85
days
  Abdominal pain (n=86, 85) | 0.227 (0.2500) | 0.216 (0.2251)
  Mild abdominal pain (n=58, 57) | 0.302 (0.2440) | 0.308 (0.2199)
  Moderate abdominal pain (n=37, 39) | 0.434 (0.2496) | 0.374 (0.2269)
  Severe abdominal pain (n=14, 12) | 0.429 (0.2646) | 0.400 (0.2741)
  Flatulence (n=86, 85) | 0.365 (0.3215) | 0.329 (0.3290)
  Mild flatulence (n=67, 61) | 0.467 (0.2912) | 0.459 (0.3018)
  Moderate flatulence (n=35, 40) | 0.351 (0.2649) | 0.577 (0.2806)
  Severe flatulence (n=20, 13) | 0.616 (0.2959) | 0.554 (0.1968)

7. Secondary Outcome: Percentage of Participants With Abdominal Distension
Description: Abdominal distension is a sense of increased abdominal pressure by the participant that involves an actual measurable change in the circumference of a participant's abdomen on physical examination. Percentage of participants with abdominal distension was calculated for each treatment period (Day 1 to Day 15).
Time Frame: Day 1 up to Day 15 in first and second treatment periods
Population: ITT population included all randomized participants. Here, 'N' specifies number of participants who had abdominal distension assessment at screening and end of specified treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Panzytrat® | Kreon®
Number analyzed (Participants) | 86 | 85
percentage of participants | 12.8 | 11.8

8. Secondary Outcome: Percent Coefficient of Fat Absorption (CFA) Based on Concomitant Use of Proton Pump Inhibitors (PPIs)
Description: Percent CFA was calculated as ([fat intake - fat excretion]/fat intake)*100, determined in the stools which were collected over a 3-day period (Day 12 to morning of Day 15) during each treatment period. Least squares mean percent (%) CFA was calculated for Day 12 to Day 15 in first and second treatment periods. Percent CFA was based on log transformed data. Percent CFA was calculated separately for participants who used and did not use acid suppressing therapy (PPIs) during the study.
Time Frame: Day 12 up to Day 15 in first and second treatment periods
Population: Per protocol population. Here, 'n' specifies number of participants who were evaluable for specific categories for each arm group, respectively.
Measure: Least Squares Mean (Standard Error); unit: percent CFA
Arm/Group | Panzytrat® | Kreon®
Number analyzed (Participants) | 38 | 38
percent CFA
  PPIs used (n=7, 7) | 79.66 (1.071) | 94.29 (1.071)
  PPIs not used (n=31, 31) | 80.89 (1.037) | 79.24 (1.037)

9. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) or Serious Adverse Events (SAEs)
Description: An AE was defined as any untoward medical occurrence regardless of its causal relationship to study drug. A TEAE was defined as any event not present prior to exposure to study drug or any event already present that worsens in either intensity or frequency following exposure to test drug. A SAE was defined as any event that results in death, is immediately life threatening, requires hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, or is a congenital anomaly/birth defect or is assessed as medically important.
Time Frame: Baseline up to 30 days after last dose
Population: Safety population included all randomized participants who received at least 1 dose of study medication. Here, 'N' (number of participants analyzed) specifies number of participants who were evaluable for this measure.
Measure: Number; unit: participants
Arm/Group | Panzytrat® | Kreon®
Number analyzed (Participants) | 86 | 85
participants
  AEs | 32 | 20
  SAEs | 0 | 0

10. Secondary Outcome: Nutritional Status as Assessed by Body Weight
Description: Mean body weight was calculated at end of treatment (within 3 days after Day 15 of first and second treatment periods).
Time Frame: Baseline, end of treatment (within 3 days after Day 15 of first and second treatment periods) or early discontinuation
Population: Safety population included all randomized participants who received at least 1 dose of study drug. Here, 'N' specifies number of participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Panzytrat® | Kreon®
Number analyzed (Participants) | 86 | 85
kg
  Baseline | 40.82 (16.001) | 41.43 (15.861)
  End of treatment | 41.22 (15.999) | 41.88 (15.886)

11. Secondary Outcome: Nutritional Status as Assessed by Body Mass Index (BMI)
Description: Nutritional status of participants was assessed by determining their BMI. BMI was calculated by dividing body weight (kg) by square of height in meter (m). Mean BMI was calculated at end of treatment (within 3 days after Day 15 of first and second treatment periods).
Time Frame: Baseline, end of treatment (within 3 days after Day 15 of first and second treatment periods) or early discontinuation
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Panzytrat® | Kreon®
Number analyzed (Participants) | 85 | 85
kg/m^2
  Baseline | 17.84 (3.296) | 17.90 (3.264)
  End of treatment | 17.94 (3.244) | 18.01 (3.240)

12. Secondary Outcome: Nutritional Status as Assessed by Electrolytes Level
Description: Nutritional status of participants was assessed by determining their electrolytes (sodium, potassium and chloride) level. Mean electrolytes level was calculated at end of treatment (within 3 days after Day 15 of first and second treatment periods).
Time Frame: Baseline, end of treatment (within 3 days after Day 15 of first and second treatment periods) or early discontinuation
Population: Safety population included all randomized participants who received at least 1 dose of study drug. Here, 'N' specifies number of participants who were evaluable for this outcome measure and 'n' specifies number of participants who were evaluable for specific categories at each time point for each arm group, respectively.
Measure: Mean (Standard Deviation); unit: millimole/L (mmol/L)
Groups:
- Kreon®, First, Then Panzytrat®: Kreon® 25,000 capsule orally daily at a stabilized dose, as per investigator's discretion, for 14 days in first treatment period followed by Panzytrat® 25,000 capsule orally daily at a stabilized dose, as per investigator's discretion, for 14 days in second treatment period. Stabilized dose for a participant was the optimal dose determined during a qualification phase that preceded the first treatment period and was based upon the participant's usual lipase and lipid intake and total dose was not to exceed 10,000 Ph.Eur. units lipase/kg body weight/day.
Arm/Group | Panzytrat® First, Then Kreon® | Kreon®, First, Then Panzytrat®
Number analyzed (Participants) | 42 | 43
millimole/L (mmol/L)
  Sodium: Baseline (n=42, 43) | 138.41 (3.026) | 138.54 (3.356)
  Sodium: End of treatment (n=42, 43) | 139.11 (2.350) | 139.07 (2.466)
  Potassium: Baseline (n=42, 42) | 4.441 (0.4799) | 4.371 (0.3721)
  Potassium: End of treatment (n=42, 42) | 4.322 (0.4113) | 4.344 (0.3506)
  Chloride: Baseline (n=38, 40) | 102.08 (3.436) | 101.40 (3.193)
  Chloride: End of treatment (n=38, 40) | 102.13 (2.796) | 102.18 (2.541)

13. Secondary Outcome: Nutritional Status as Assessed by Albumin, Serum Transferrin and Hemoglobin Level
Description: Nutritional status of participants was assessed by determining their albumin, serum transferrin and hemoglobin level. Mean albumin, serum transferrin and hemoglobin level was calculated at end of treatment (within 3 days after Day 15 of first and second treatment periods).
Time Frame: Baseline, end of treatment (within 3 days after Day 15 of first and second treatment periods) or early discontinuation
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: gram/L (g/L)
Arm/Group | Panzytrat® First, Then Kreon® | Kreon® First, Then Panzytrat®
Number analyzed (Participants) | 42 | 42
gram/L (g/L)
  Albumin: Baseline (n=41, 42) | 40.553 (11.3568) | 37.995 (14.8405)
  Albumin: End of treatment (n=41, 42) | 40.785 (11.1893) | 37.991 (14.9636)
  Serum transferrin: Baseline (n=40, 41) | 2.877 (0.9769) | 2.618 (1.1857)
  Serum transferrin: End of treatment (n=40, 41) | 2.916 (0.9416) | 2.626 (1.1618)
  Hemoglobin: Baseline (n=42, 42) | 137.337 (11.7570) | 141.118 (11.4577)
  Hemoglobin: End of treatment (n=42, 42) | 137.935 (11.4543) | 141.263 (11.4412)

14. Secondary Outcome: Nutritional Status as Assessed by Hematocrit Level
Description: Nutritional status of participants was assessed by determining their hematocrit level. Mean hematocrit level was calculated at end of treatment (within 3 days after Day 15 of first and second treatment periods).
Time Frame: Baseline, end of treatment (within 3 days after Day 15 of first and second treatment periods) or early discontinuation
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: proportion of hematocrit
Arm/Group | Panzytrat® First, Then Kreon® | Kreon® First, Then Panzytrat®
Number analyzed (Participants) | 42 | 42
proportion of hematocrit
  Baseline | 0.408 (0.0324) | 0.417 (0.0333)
  End of treatment | 0.409 (0.0311) | 0.416 (0.0328)

ADVERSE EVENTS:
Time Frame: Baseline up to 30 days after last dose
Description: Adverse event (AE) was any untoward medical occurrence regardless of causal relationship to study drug. Serious AE was any event that resulted in death, life threatening, required or prolonged in-patient hospitalization, significant disability/incapacity, or was a congenital anomaly/birth defect. Participants at risk: Panzytrat®=86 and Kreon®=85.
Arm/Group | Panzytrat® | Kreon®
Serious Adverse Events (participants affected / at risk) | 0/86 | 0/85
Other Adverse Events (participants affected / at risk) | 32/86 | 20/85
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Panzytrat® (N=86) | Kreon® (N=85)
Flatulence (Gastrointestinal disorders) | 15 | 6
Abdominal pain (Gastrointestinal disorders) | 11 | 9
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1
Rhinitis (Infections and infestations) | 1 | 1
Gastrointestinal infection (Infections and infestations) | 1 | 0
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1
Varicella (Infections and infestations) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pyrexia (General disorders) | 2 | 2
Headache (Nervous system disorders) | 2 | 1
Pseudomonas test positive (Investigations) | 0 | 1
Vitamin A decreased (Investigations) | 1 | 0
Conjunctivitis (Eye disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Haematoma (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Restrictions vary in accordance with each agreement with the individual investigators. Sponsor will allow publication after a multi-center publication has been published or after an agreed period of time if no such multi-center publication is submitted for publication. Sponsor can ask that Sponsor's confidential information be removed from any publication and can defer publication for a period of time to allow for Sponsor to obtain patent or other intellectual property right protection.